CLINICAL TRIAL: NCT06725355
Title: A Bioequivalence Study to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety After Administration of IN-R00002 and IN-G00002 in Healthy Adult Volunteers
Brief Title: To Compare the Pharmacokinetics and Safety After a Single Dose Administration of IN-G00002 and IN-R00002 in Healthy Adult Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_LXA_101
Record Dates: First submitted 2024-11-25; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Experimental): R->T R: IN-R00002 T: IN-G00002
  Interventions: Drug: IN-R00002; Drug: IN-G00002
- Sequence B (Experimental): T->R R: IN-R00002 T: IN-G00002
  Interventions: Drug: IN-R00002; Drug: IN-G00002

INTERVENTIONS:
Drug: IN-R00002 — Single administration of IN-R00002 60mg
Drug: IN-G00002 — Single administration of IN-G00002 60mg

SUMMARY:
To compare the pharmacokinetics and safety after a single dose administration of IN-G00002 and IN-R00002 in healthy adult volunteers

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, crossover study

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged ≥ 19 years at screening
* Body weight > 60kg and Body mass index (BMI) in the range of 18.0 and 30.0 kg/㎡
* Subjects who do not have congenital or chronic diseases requiring treatment and have no pathological symptoms or findings as a result of physical examination
* Determined by the investigator to be eligible for study participation based on the results of screening tests (clinical laboratory tests, vital signs, physical examination, 12-lead ECG) conducted according to the IP characteristics
* Subjects who decided to participate in the study and signed informed consent form voluntarily after receiving detailed explanation of the study and fully understanding

Exclusion Criteria:

* Subjects who have taken the drug which can induce or inhibit drug metabolism enzyme within 4 weeks prior to the 1st IP administration
* Subjects who have participated in any other clinical study or bioequivalnece study within 6 months prior to the 1st IP administration
* Subjects who have donated whole blood within 8 weeks prior to the 1st IP administration or have donated blood components or received transfusion within 2 weeks prior to the 1st IP administration
* Pregnant(positive urine HCG) or breastfeeding women if female
* Subject who have continued drink of alcohol within 1 month prior to the 1st IP administration (female: > 14 glasses per week, male > 21 glasses per week)
* Subjects with a presence and a history of surgery or gastrointestinal diseases which might significantly change absorption of medicines
* Pregnant(positive urine HCG) or breastfeeding women if female
* Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects or spouses (or partners) are unable to use an effective method of contraception (e.g., correctly placed intrauterine device, sterilization surgery (vasectomy, tubal ligation, etc.), barrier method (spermicide and condom, a concomitant use of contraceptive diaphragm, vaginal sponge or cervical cap)), throughout the study
* Subjects who are judged ineligible for the clinical study by the investigator due to reasons other than the above inclusion/exclusion criteria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
PK parameter | Up to Day 2
  AUClast of Edoxaban
PK parameter | Up to Day 2
  Cmax of Edoxaban

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Clinical Trial Center, Siheung, South Korea